CLINICAL TRIAL: NCT06122467
Title: A Single Group Study to Evaluate the Efficacy of a Cosmetic Product Line on Acne Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menning Labs (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20365
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group: EQ Product Line (Experimental): The following regimen should be completed in both the morning and the evening. The order of use is:
  Cleanser Gel Moisturizer.
  Interventions: Other: EQ Exfoliating Cleanser; Other: EQ Gel; Other: EQ Moisturizer

INTERVENTIONS:
Other: EQ Exfoliating Cleanser — Product contains: Purified water, disodium laureth sulfosuccinate, coco betaine, decyl glucoside, Juglans regia (walnut) shells, PEG-40 hydrogenated castor oil, sodium cocoyl isethionate disodium cocoyl glutamate, ethoxydiglycol, xanthan gum, Root Blend Preservative (hexylene glycol, caprylyl glycol, Wasabia japonica (wasabi) root extract, Zingiber officinale (ginger) root extract, Allium sativum (garlic) bulb extract), Aloe barbadensis (aloe vera) leaf juice concentrate (Aloe barbadensis leaf juice, potassium sorbate, sodium benzoate, citric acid).
Other: EQ Gel — Product contains: Purified water, witch hazel (containing 14% grain alcohol), PEG-40 hydrogenated castor oil, ethoxydiglycol, xanthan gum, Root Blend Preservative (hexylene glycol, caprylyl glycol, Wasabia japonica (wasabi) root extract, Zingiber officinale (ginger) root extract, Allium sativum (garlic) bulb extract), xanthan gum.
Other: EQ Moisturizer — Product contains: Purified water, glycerin, dicaprylyl carbonate, cetyl alcohol, glyceryl stearate citrate, squalane, PEG-40 hydrogenated castor oil, caprylic/capric triglycerides, stearic acid, jojoba oil, phenoxyethanol SA (phenoxyethanol, caprylyl glycol, sorbic acid), ethoxydiglycol, Root Blend Preservative (hexylene glycol, caprylyl glycol, Wasabia japonica (wasabi) root extract, Zingiber officinale (ginger) root extract, Allium sativum (garlic) bulb extract), allantoin, sodium carbomer.

SUMMARY:
This twelve-week trial will examine the effectiveness of a Menning Labs EQ Product Line acne product. Participants will use the exfoliating cleanser, cream, and gel daily for 8 weeks. Participants will complete questionnaires at Baseline, Day 1, Day 3, Day 7, Day 28, Day 42, and Day 56. Participants will also provide before-and-after photos at Baseline, Day 7, and Day 42, as well as undergo expert skin grading at Baseline and Day 42. The questionnaire on Day 56 will mark the conclusion of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Be aged between 18-45.
* Anyone who has acne prone skin and a history of recurring acne.
* Has visible acne at enrollment.
* Anyone who is generally healthy - does not live with any uncontrolled chronic disease.
* Have a digital camera or smartphone to take photos of the face.

Exclusion Criteria:

* Anyone with pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Anyone currently using a prescription skin product.
* Anyone who is unwilling to stop using the current acne supplements they are taking.
* Anyone with known severe allergic reactions.
* Any women who are pregnant, breastfeeding or attempting to become pregnant.
* Anyone unwilling to follow the study protocol.
* Anyone who identifies as having sensitive skin.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the appearance of facial skin acne. [Timeframe: Baseline to Day 56] | 56 days
  Assessed via expert skin grading of baseline and endline photos conducted by a board-certified dermatologist.
  Study-specific surveys using a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe"). Surveys will be completed independently by study participants.
Changes in skin clarity i.e. reduction in acne or associated blemishes. [Timeframe: Baseline to Day 56] | 56 days
  Assessed via expert skin grading of baseline and endline photos conducted by a board-certified dermatologist.
  Study-specific surveys using a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe"). Surveys will be completed independently by study participants.

SECONDARY OUTCOMES:
Changes in overall skin health. [Timeframe: Baseline to Day 56] | 56 days
  Assessed via expert skin grading of baseline and endline photos conducted by a board-certified dermatologist.
  Study-specific surveys using a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe"). Surveys will be completed independently by study participants.
Changes in skin texture. [Timeframe: Baseline to Day 56] | 56 days
  Assessed via expert skin grading of baseline and endline photos conducted by a board-certified dermatologist.
  Study-specific surveys using a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe"). Surveys will be completed independently by study participants.
Changes in facial skin irritation. [Timeframe: Baseline to Day 56] | 56 days
  Surveys will be completed independently by study participants. Study-specific surveys using a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in skin redness. [Timeframe: Baseline to Day 56] | 56 days
  Assessed via expert skin grading of baseline and endline photos conducted by a board-certified dermatologist.
  Study-specific surveys using a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe"). Surveys will be completed independently by study participants.
Changes in skin smoothness. [Timeframe: Baseline to Day 56] | 56 days
  Assessed by surveys completed independently by study participants. Study-specific surveys using a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No